CLINICAL TRIAL: NCT00997607
Title: A Phase IB Study to Evaluate the Safety and Immunogenicity of an Ebola DNA Plasmid Vaccine, VRC-EBODNA023-00-VP, and a Marburg DNA Plasmid Vaccine, VRC-MARDNA025-00-VP, in Healthy Adults in Kampala, Uganda
Brief Title: Evaluating an Ebola and a Marburg Vaccine in Uganda
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 247
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Ebola Virus Disease; Marburg Virus Disease
Keywords: Vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Marburg Virus Disease | interventions — Ebola Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ebola vaccine only (Experimental): Participants will receive only the Ebola vaccine or a placebo injection.
  Interventions: Biological: Ebola vaccine; Other: Placebo injection
- Marburg vaccine only (Experimental): Participants will receive only the Marburg vaccine or a placebo injection.
  Interventions: Biological: Marburg vaccine; Other: Placebo injection
- Ebola and Marburg vaccine (Experimental): Participants will receive both the Ebola and Marburg vaccines, one in each arm or placebo injections.
  Interventions: Biological: Ebola vaccine; Biological: Marburg vaccine; Other: Placebo injection

INTERVENTIONS:
Biological: Ebola vaccine — 4 mg of Ebola DNA plasmid vaccine, VRC-EBODNA023-00-VP, delivered via intramuscular injection on Weeks 0, 4, and 8
  Arms: Ebola and Marburg vaccine; Ebola vaccine only
Biological: Marburg vaccine — 4 mg of Marburg DNA plasmid vaccine, VRC-MARDNA025-00-VP, delivered via intramuscular injection on Weeks 0, 4, and 8
  Arms: Ebola and Marburg vaccine; Marburg vaccine only
Other: Placebo injection — 4 mg of saline injection delivered at Weeks 0, 4, and 8

SUMMARY:
This study will test two new vaccines, one for Ebola and one for Marburg virus, to see if they are safe, if they have side effects, and if they create an immune response in people who receive them.

DETAILED DESCRIPTION:
The Ebola and Marburg viruses are both filoviruses known to induce hemorrhagic fever-a set of symptoms characterized by sudden onset, aching, fever, and bleeding in the internal organs. Both filoviruses are associated with high mortality rates, and the Centers for Disease Control (CDC) lists them as Category A bioterrorism agents because of their potential for a major public health impact. Vaccines for both viruses are under development using a prime-boost strategy that involves multiple injections over a period of time to confer long-lasting immunity. Preliminary research supports the vaccines' safety. This study will test these experimental vaccines for the Ebola and Marburg viruses, first administered separately and then together, to ensure they are safe and do not have side effects.

Participation in this study will entail 11 study visits over 2 years. The study will have two parts, to be completed sequentially, and three groups. In part one, participants will be randomly assigned to the first group, which will receive the experimental Ebola DNA vaccine, or the second group, which will receive the experimental Marburg DNA vaccine. In part two, the third group will receive both the Ebola and the Marburg vaccines, one shot in each arm. One fifth of the participants in each group will be controls and receive placebo injections. All vaccines and placebos will be delivered via an intramuscular injection at three time points: at study entry, after 4 weeks, and after 8 weeks.

Participants will complete study assessments at 12 points in time: at baseline and at Weeks 2, 4, 6, 8, 10, 12, 24, 32, 52, 78, and 104. At each assessment, changes in health and medications will be recorded and blood will be drawn. Participants will also complete a diary card daily for 5 days after receiving each injection. In it, they will record their temperature and any skin changes at the injection site.

ELIGIBILITY:
Inclusion Criteria:

* Available for clinical follow-up through Week 104
* Willing to have photo taken for identification purposes
* Willing to be taken home at enrollment visit and allow home visits if appointments are not kept
* Completes an Assessment of Understanding (AoU) prior to enrollment by answering 9 out of 10 questions at least once in 3 attempts
* In good general health without clinically significant medical history
* Has a physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment
* Female participants of reproductive potential must have a negative result on a human choriogonadotropin (β-HCG) pregnancy test
* Female participants must either be incapable of becoming pregnant or agree to take appropriate precautions that pregnancy will not occur during the first 24 weeks of the study

Exclusion Criteria:

* Pregnant, breast-feeding, or planning to become pregnant during the first 24 weeks after enrollment
* History of Ebola or Marburg virus exposure
* Occupational health risk of exposure to the Ebola or Marburg virus known to be higher than that of the general population
* Has received any of the following substances:

  * Investigational Ebola or Marburg vaccine in a prior clinical trial
  * Blood products within 120 days prior to HIV screening
  * Immunoglobulin within 60 days of prior to HIV screening
  * Live attenuated vaccines within 30 days prior to initial study vaccine administration
  * Investigational research agents within 30 days prior to initial study vaccine administration
  * Medically indicated subunit or killed vaccines (such as influenza, pneumococcal, or allergy treatment with antigen injections) within 14 days of study vaccine administration
  * Current anti-tuberculosis prophylaxis or therapy
  * Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within 12 weeks of enrollment, except in the following cases: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroids for a non-chronic condition (based on investigator clinical judgement) at least 2 weeks prior to enrollment in this study
* History of serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain
* Presence of idiopathic urticaria within the past 2 years
* History of autoimmune disease or immunodeficiency
* History of unstable asthma; asthma that required emergent care, urgent care, hospitalization or intubation during the past 2 years; or asthma that requires the use of oral or parenteral corticosteroids
* History of diabetes mellitus (type I or II), with the exception of a history of gestational diabetes
* History of thyroidectomy or thyroid disease that required medication within the past 12 months
* History of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema
* History of hypertension that is not well controlled by medication or blood pressure that is more than 145/95 mm Hg at enrollment
* Presence of a bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions), significant bruising or bleeding difficulties with intramuscular injections or blood draws, or routine use of anticoagulant medications
* Presence of active malignancy, treated malignancy for which there is not reasonable assurance of sustained cure, or malignancy that is likely to recur during the period of the study
* History of a seizure or seizure disorder
* Asplenia, functional asplenia, or any condition resulting in the absence or removal of the spleen
* Allergic reaction to aminoglycoside antibiotics
* Presence of a psychiatric condition that precludes compliance with the protocol
* History of psychoses, bipolar disorder, disorder requiring lithium, or suicide plan or attempt within 5 years prior to enrollment
* Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent
* Evidence of syphilis based on history, exam, and rapid plasma reagin (RPR) test results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety of Ebola vaccine, as seen in local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and serious adverse experiences | Measured at 11 or more visits over 2 years
Safety of Marburg vaccine, as seen in local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and serious adverse experiences | Measured at 11 or more visits over 2 years

SECONDARY OUTCOMES:
Immunogenicity of Ebola vaccine, as seen in ELISA antigen-specific assays for antibodies, intracellular cytokine staining (ICS) assay, and an ELISPOT antigen-specific assay for T cell responses | Measured at baseline and Week 12
Immunogenicity of Marburg vaccine, as seen in ELISA antigen-specific assays for antibodies, intracellular cytokine staining (ICS) assay, and an ELISPOT antigen-specific assay for T cell responses | Measured at baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Kibuuka, MBChB, MMed, MPH, Principal Investigator — Makerere University
Locations (1):
- Makerere University Walter Reed Project (MUWRP) clinic, Kampala, Uganda

REFERENCES:
- [Derived] Kibuuka H, Berkowitz NM, Millard M, Enama ME, Tindikahwa A, Sekiziyivu AB, Costner P, Sitar S, Glover D, Hu Z, Joshi G, Stanley D, Kunchai M, Eller LA, Bailer RT, Koup RA, Nabel GJ, Mascola JR, Sullivan NJ, Graham BS, Roederer M, Michael NL, Robb ML, Ledgerwood JE; RV 247 Study Team. Safety and immunogenicity of Ebola virus and Marburg virus glycoprotein DNA vaccines assessed separately and concomitantly in healthy Ugandan adults: a phase 1b, randomised, double-blind, placebo-controlled clinical trial. Lancet. 2015 Apr 18;385(9977):1545-54. doi: 10.1016/S0140-6736(14)62385-0. Epub 2014 Dec 23. PMID 25540891